CLINICAL TRIAL: NCT04531410
Title: Double-blind Randomized Controlled Study of Linoleic Acid Supplementation for 1 Year in Patients With Cystic Fibrosis - Influence on Clinical Status and Metabolism
Brief Title: NETwork of Linoleic Acid Supplementation in Cystic Fibrosis
Acronym: NETLACF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: European Society of Pediatric Gastroenterology, Hepatology and Nutrition (Other)
Responsible Party: Principal Investigator, Birgitta Strandvik, MD, PhD, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-02871
Record Dates: First submitted 2020-08-18; First posted 2020-08-28 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Cystic Fibrosis
Keywords: arachidonic acid,; lipid mediators; cytokines; growth; pulmonary function; IGF-1; resting energy expenditure; docosahexaenoic acid
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Parallel, double blind, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The supplement only differ by colour on capsulae, no labelling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linoleic (Experimental): Linoleic acid 13 g and 600 mg algal docosahexaenoic acid (DHA)
  Interventions: Dietary Supplement: linoleic acid supplementation
- Oleic (Active Comparator): Oleic acid 13 g and 600 algal DHA
  Interventions: Dietary Supplement: oleic acid supplementation

INTERVENTIONS:
Dietary Supplement: linoleic acid supplementation — Oils given daily at morning meal with extra enzymes
  Arms: Linoleic
Dietary Supplement: oleic acid supplementation — Oils given at morning meal with extra enzymes
  Arms: Oleic

SUMMARY:
Undernutrition is a common problem in patients with cystic fibrosis (CF) despite international consensus that the patients shall be given 120-200% of energy recommendations. Studies imply that one problem might be that the patients are not compensated for the essential fatty acid deficiency (linoleic acid, LA), which is well known in these patients. This deficiency is shown not to be due to fat malabsorption, but related to an increased turnover of arachidonic acid, a transformation product of LA. This abnormality is related to mutations associated with a more severe clinical phenotype. The most common and typical symptom of LA deficiency is poor growth. Studies in animals have further indicated that many of the symptoms in CF are related to the deficiency. A series of recent prospective studies from Wisconsin corroborate the importance of LA for growth. In Sweden LA has been supplemented to most patients since the late 70´, and the condition of patients have been among the leading in the world regarding growth, pulmonary function and survival. Short-term studies have shown better effect of LA supplementation compared to similar supply of energy without including extra LA. There are few long-term studies, performed before the gene was identified, giving very heterogeneous patient groups in regard to genotype, but with some positive results on growth and physiology. It´s of interest that modern personalized extremely expensive therapy with correctors and potentiators for Cystic Fibrosis Transmembrane Conductance Regulator may influence lipid metabolism. LA might thus tentatively be a cheap adjuvant to this modern therapy, but this has to be specially studied.

The aim of the study is to find if there are differences in clinical and metabolic outcome between two groups, blindly given similar amount of extra calories, in one group consisting of linoleic acid.The benefit for the patients would be great if the expected positive effect can be proved in the planned study. The treatment will be cheap and without adverse effects. From socioeconomic point of view is would be a great advantage.

DETAILED DESCRIPTION:
Two group of matched children with CF were randomized to two type of oils given 20 g oil and 600 mg DHA daily for one year and anthropometry, pulmonary function, biochemistry, resting energy expenditure, lipid mediators, inflammatory and intestinal markers were studied at start and at 6 months and 1 year. Dietary intake was controlled and life quality recording at start and end of study.

ELIGIBILITY:
Inclusion Criteria:

* Two mutations related to severe clinical status such as dF508, or other stop mutations or class II mutations. Severe status includes pancreatic insufficiency

Exclusion Criteria:

* Liver cirrhosis and/or portal hypertension, transplantation or on transplantation list, intake of lipid supplements the latest 2 months

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Try to have similar number of participants of the same sex and age for randomization
Enrollment: 50 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Growth | 1 year
  change in BMI, standard deviation score (SDS)
Weight | 1 year
  change in SDS body weight
Height | 1 year
  change in SDS height

SECONDARY OUTCOMES:
Pulmonary function | 1 year
  change in forced expiratory volume in one second (FEV1 % of predicted)
Quality of life, the patient experience of well being | 1 year
  Questionaire about health, physical activity, well being (8 items), CFQ-child + CFQ- parents (higher rates are better) The score changes are analysed.The CFQ considers the physical, image, digestive, respiratory, emotional, social, food, treatment, vitality, health, social role and weight domains. Each domain has a score and its sum generates the total score, whose values can vary from 0 to 100 The scores will also be related to measurements.

OTHER OUTCOMES:
Lipid mediators | 1 year
  change in lipid mediators in blood and urine, ion trap- Mass Spectrometry, picoMol (> 150 products of both the n-6 and n-3 series)
Clinical infectious status | 1 year
  change in number exacerbations compare to previous year,
Influence on sodium status | 1 year
  change in Sodium in sweat test, mol/L and urine (fractional sodium excretion)
Inflammatory markers | 1 year
  change in Cytokines, Proximity extension assays (PEA proteomics) picogram/ml
Metabolic marker | 1 year
  Change in serum insulin growth factor -1 (IGF-1, nanogram/ml)
Energy metabolism | 1 year
  Change in resting energy expenditure (REE/kg body weight)
Bone mineral density | 1 year
  Change in total bone mineral density by dual x-ray absorptiometry (DXA), gram/cm^2
Oral glucose tolerance | 1 year
  Measure of glucose and insuline after oral glucose loading

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw Walkowiak, MD,PhD, Principal Investigator — University of Poznan, CF center, Poland; Carla Colombo, MD,PhD, Principal Investigator — University of Milan, CF center, Italy; Egil Bakkeheim, MD, PhD, Principal Investigator — University of Oslo, CF center, Norway; Raffaele Badolato, MD, PhD, Principal Investigator — University of Brescia, CF center, Italy; Christine Rönne-Hansen, Md, PhD, Principal Investigator — Lund University, CF center, Sweden
Locations (3):
- Università degli Studi di Milan, Milan, Italy
- Norwegian Resourse Center for Cystic Fibrosis, Oslo University Hospital, Oslo, Norway
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No
The results will be anonymous and reported to peer review journals for publication. Beside the local PIs there will be other local staff involved and for the analyses also co-workers as shown in the study protocol which will be attached for review.

REFERENCES:
- [Background] Strandvik B. Fatty acid metabolism in cystic fibrosis. Prostaglandins Leukot Essent Fatty Acids. 2010 Sep;83(3):121-9. doi: 10.1016/j.plefa.2010.07.002. Epub 2010 Jul 31. PMID 20673710
- [Background] Wheelock CE, Strandvik B. Abnormal n-6 fatty acid metabolism in cystic fibrosis contributes to pulmonary symptoms. Prostaglandins Leukot Essent Fatty Acids. 2020 Sep;160:102156. doi: 10.1016/j.plefa.2020.102156. Epub 2020 Jun 26. PMID 32750662
- [Background] Strandvik B. Is the ENaC Dysregulation in CF an Effect of Protein-Lipid Interaction in the Membranes? Int J Mol Sci. 2021 Mar 8;22(5):2739. doi: 10.3390/ijms22052739. PMID 33800499
- [Background] Strandvik B. Nutrition in Cystic Fibrosis-Some Notes on the Fat Recommendations. Nutrients. 2022 Feb 18;14(4):853. doi: 10.3390/nu14040853. PMID 35215502

DOCUMENTS (5):
  • Study Protocol (2024-11-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT04531410/Prot_003.pdf
  • Statistical Analysis Plan (2024-11-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT04531410/SAP_004.pdf
  • Informed Consent Form: Ethical approvement (2024-11-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT04531410/ICF_005.pdf
  • Informed Consent Form: Patients info consent (2024-11-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT04531410/ICF_006.pdf
  • Informed Consent Form: Patient information Parents (2024-11-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT04531410/ICF_007.pdf